CLINICAL TRIAL: NCT02372019
Title: Augmenting Interpretative Cognitive Bias Modification Using Memory Reconsolidation Updating
Brief Title: Augmentation Study of A Computerized Treatment for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-11-0009
Record Dates: First submitted 2015-02-10; First posted 2015-02-26 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Social Phobia; Reconsolidation; Cognitive Bias Modification; Interpretation Bias
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBM With Active Fear Reactivation (Experimental)
  Interventions: Behavioral: CBM With Active Fear Reactivation
- CBM With Inert Fear Reactivation (Active Comparator)
  Interventions: Behavioral: CBM With Inert Fear Reactivation
- Inert CBM With Inert Fear Reactivation (Placebo Comparator)
  Interventions: Behavioral: Inert CBM With Inert Fear Reactivation

INTERVENTIONS:
Behavioral: CBM With Active Fear Reactivation — Participants will undergo a fear reactivation trial, which involves giving a one-minute impromptu speech after only 30 seconds of preparation time. 10 minutes afterwards, they will be given CBM for interpretation bias. Training will involve 84 social scenario vignettes, with 70 resolving positively, 7 resolving negatively, and 7 resolving neutrally. This training takes places during the "memory reconsolidation window" that opens after fear reactivation, during which time the fear memory is in a labile state and thus more amenable to rewriting.
  Arms: CBM With Active Fear Reactivation
Behavioral: CBM With Inert Fear Reactivation — Participants will undergo a fear reactivation trial, which involves giving a one-minute impromptu speech after only 30 seconds of preparation time. 12 to 36 hours afterwards, they will be given CBM for interpretation bias. Training will involve 84 social scenario vignettes, with 70 resolving positively, 7 resolving negatively, and 7 resolving neutrally. Because this training takes places well outside of the "memory reconsolidation window" that opens shortly after fear reactivation, the reactivation is not expected to have any effect, and only serves as a control.
  Arms: CBM With Inert Fear Reactivation
Behavioral: Inert CBM With Inert Fear Reactivation — Participants will undergo a fear reactivation trial, which involves giving a one-minute impromptu speech after only 30 seconds of preparation time. 12 to 36 hours afterwards, they will be given an inert form of CBM, which should not influence the direction of interpretation bias. Training will involve 84 social scenario vignettes, with 70 resolving neutrally, 7 resolving positively, and 7 resolving negatively. Because the CBM training takes places well outside of the "memory reconsolidation window" that opens after fear reactivation, the reactivation is not expected to have any effect, and the inert CBM training is not expected to have any effect either. This condition only serves as a control for the other two conditions.
  Arms: Inert CBM With Inert Fear Reactivation

SUMMARY:
The purpose of this study is to determine whether briefly reactivating a fear memory 10 minutes prior to administering a social anxiety treatment will enhance the durability of treatment effects.

DETAILED DESCRIPTION:
This study examines whether cognitive bias modification of interpretation (CBM-I) for socially anxious individuals can be augmented with the inclusion of a fear memory reactivation prior to administration of CBM. To date, CBM-I generally involves presenting participants with short vignettes that have ambiguous meaning. The ambiguity is resolved by having the subject complete a word stem at the conclusion of the paragraph, resolving the ambiguity in a positive/negative/neutral fashion. CBM attempts to retrain the tendency for socially phobic individuals to adopt negative interpretations of ambiguous events by repeatedly presenting trials resolving in a positive fashion. An inert control can be administered by having the majority of CBM trials resolve in a neutral fashion, without having the vignette end in either a positive or negative fashion.

Reactivating a fear memory, followed by a short break, purportedly opens a window of several hours during which the fear memory is rendered labile, and so CBM given during this time should show greater durability of effects. However, manipulations given outside of this timeframe will presumably have no increased effects. Individuals exhibiting clinical levels of social anxiety, as measured with the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria, will be randomly assigned to one of three conditions: (1) fear reactivation administered 10 minutes prior to CBM, (2) fear reactivation administered 12-36 hours prior to CBM, and (3) fear reactivation administered 12-36 hours prior to an inert form of CBM. A variety of measures measuring anxiety, interpretation bias, and cognitions will be repeatedly assessed across the study, including at pretreatment, post treatment, and at one and two week follow up. Additionally, several potential moderators of treatment outcome will be assessed prior to engaging in treatment. At two week follow up, participants will also be given a speech stressor task to determine its effect on subsequent interpretation bias.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Score of 30 or above on LSAS
* Score of 1.4 or greater on ASSIQ

Exclusion Criteria:

* Receiving any form of anxiety medication or psychotherapy for anxiety during the past 3 months
* Scoring above a "1" on item 9 of the BDI-II (presence of serious suicidal ideation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Liebowitz Social Anxiety Scale (LSAS) at 24 Hours | pretreatment, 24-hour follow up
  The LSAS is a commonly used measure of social anxiety that measures fear as well as avoidance behaviors concerning social interactions. The study will use a computerized, self-report version of the LSAS, which has demonstrated little deviation from clinician-administered LSAS scores.
Change From Baseline in Liebowitz Social Anxiety Scale (LSAS) at 1 Week | pre-treatment, 1-week follow up
  The LSAS is a commonly used measure of social anxiety that measures fear as well as avoidance behaviors concerning social interactions. The study will use a computerized, self-report version of the LSAS, which has demonstrated little deviation from clinician-administered LSAS scores.
Change From Baseline in Liebowitz Social Anxiety Scale (LSAS) at 2 Weeks | pre-treatment, 2-week follow up
  The LSAS is a commonly used measure of social anxiety that measures fear as well as avoidance behaviors concerning social interactions. The study will use a computerized, self-report version of the LSAS, which has demonstrated little deviation from clinician-administered LSAS scores.
Change From Baseline in Brief Fear of Negative Evaluation Scale (BFNE) at 24 Hours | pretreatment, 24-hour follow up
  The 12-item, self-report Brief Fear of Negative Evaluation Scale measures fear of negative evaluation by others, which is a distinguishing characteristic of social anxiety. The scale is derived from the original 30-item Fear of Negative Evaluation measurement.
Change From Baseline in Brief Fear of Negative Evaluation Scale (BFNE) at 1 Week | pretreatment, 1-week follow up
  The 12-item, self-report Brief Fear of Negative Evaluation Scale measures fear of negative evaluation by others, which is a distinguishing characteristic of social anxiety. The scale is derived from the original 30-item Fear of Negative Evaluation measurement.
Change From Baseline in Brief Fear of Negative Evaluation Scale (BFNE) at 2 Weeks | pretreatment, 2-week follow up
  The 12-item, self-report Brief Fear of Negative Evaluation Scale measures fear of negative evaluation by others, which is a distinguishing characteristic of social anxiety. The scale is derived from the original 30-item Fear of Negative Evaluation measurement.
Change From Baseline in Appraisal of Social Concerns Scale (ASC) at 24 Hours | pretreatment, 24-hour follow up
  The ASC is a 20-item self-report questionnaire that focuses on cognitions present in socially anxious patients. It measures concerns about negative evaluation, observable symptoms, and perceived social helplessness.
Change From Baseline in Appraisal of Social Concerns Scale (ASC) at 1 Week | pretreatment, 1-week follow up
  The ASC is a 20-item self-report questionnaire that focuses on cognitions present in socially anxious patients. It measures concerns about negative evaluation, observable symptoms, and perceived social helplessness.
Change From Baseline in Appraisal of Social Concerns Scale (ASC) at 2 Weeks | pretreatment, 2-week follow up
  The ASC is a 20-item self-report questionnaire that focuses on cognitions present in socially anxious patients. It measures concerns about negative evaluation, observable symptoms, and perceived social helplessness.

SECONDARY OUTCOMES:
Word Sentence Association Paradigm (WSAP) | pretreatment (assessed twice: before & after fear retrieval), post-treatment (within 30 minutes following CBM administration), 1-week follow up, 2-week follow up (assessed twice at 2-week follow up: before and after a speech task stressor)
  This measure of interpretation bias involves a series of trials in which an ambiguous sentence describing a social situation is presented, followed by the presentation of a single word corresponding to either a threat interpretation or a benign interpretation of the sentence. The participant's task is to indicate whether the sentence and the word are related.
Ambiguous Social Scenarios Interpretation Questionnaire (ASSIQ) | pretreatment, post-treatment (within 30 minutes following CBM administration), 1-week follow up, 2-week follow up (assessed twice at 2-week follow up: before and after a speech task stressor)
  The ASSIQ is an alternative measure of interpretation bias, involving the presentation of an ambiguous social scenario, and the subsequent listing of three possible explanations corresponding to positive, neutral, and negative interpretations. Participants rate these explanations based on their likelihood of explaining the scenario. Stimuli are to be developed by the authors of the current study. In contrast to the WSAP, the ASSIQ is being used to assess more reflective aspects of interpretation bias.
Brief State-Trait Anxiety Inventory- State (BSTAI) | pretreatment (assessed 3x: before & after fear retrieval, & immediately before CBM), post treatment (within 30 minutes following CBM administration), 1-week follow up, 2-week follow up (assessed 2x at two-week follow up: before & after speech stressor)
  The BSTAI is a self-report measure comprised of six items taken from the State-Trait Anxiety Inventory, which together measure state anxiety. The BSTAI is highly correlated (r=0.93) with the full 20-item STAI. The instrument measures current state anxiety levels, but will also be administered immediately after the speech tasks to assess peak anxiety during the speech itself. During these instances, the wording of the BSTAI questions will be adapted to reflect this timing.
Perception of Speech Performance Measure (PSP) | 2-week follow up (after speech stressor task)
  This adapted 17-item measure will ask subjects to predict how others would rate the subject's own speech performance. It includes questions about both specific (voice steadiness) and global (appearance of confidence) items.
Self-Beliefs Related To Social Anxiety Scale (SBSA) | pretreatment
  The SBSA is a self-report measure that includes 15 items assessing the presence of three types of self-beliefs common in socially anxious individuals: (a) excessively high self-standards, (b) conditional self-beliefs, and (c) unconditional self-beliefs. Assessments from this scale will be examined as a potential moderator of social phobia and interpretation bias improvement.
Interpretation of Positive Events Scale (IPES) | pretreatment
  The IPES is a 13-item self-report questionnaire assessing negative interpretations of positive social events. Assessments from this scale will be examined as a potential moderator of social phobia and interpretation bias improvement.
Beck Depression Inventory-II (BDI-II) | pretreatment
  The BDI-II is a self-report scale that is among the most commonly used measures of depression. Assessments from this scale will be examined as a potential moderator of social phobia and interpretation bias improvement.
Dot Probe Task | pretreatment
  The dot probe task will be used in the current study to determine whether attentional bias moderates change in interpretation bias. The computerized paradigm involves the repeated presentation of two stimuli simultaneously, with one stimulus representing threat and the other stimulus representing safety. 500ms after stimulus onset, both stimuli are removed and one is replaced with a probe (for example, a letter would appear behind the former location of the threat stimulus or the safety stimulus). The participant's task is to determine the location of the probe. Attentional deployment prior to probe onset is inferred by response time latencies to probe location. Assessments from this task will be examined as a potential moderator of social phobia and interpretation bias improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- Laboratory for the Study of Anxiety Disorders, University of Texas at Austin, Austin, Texas, United States